CLINICAL TRIAL: NCT04412083
Title: Primary Progressive Aphasia (PPA) Tele-Savvy: A Pilot Study of an Online Intervention for Caregivers of Persons Living With PPA
Brief Title: PPA Tele-Savvy: A Pilot Study of an Online Intervention for Caregivers of Persons Living With PPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00210711
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Primary Progressive Aphasia; Caregiver Burnout
MeSH Terms: conditions — Aphasia, Primary Progressive; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPA Tele-Savvy Pilot Intervention (Other): The Tele-Savvy program is comprised of weekly, two-hour interactive classes, over seven consecutive weeks, the same duration as the proposed intervention. Tele-Savvy consists of educational instruction, video and in-class exercises that engage participants on a functional level. Course material was designed to provide informal caregivers with the knowledge, skills, and attitude needed to carry out their role as a caregiver for a person living with dementia (PLWD). Course learning objectives include: 1) introduction to dementing disorder; 2) caregiver self-care; 3) the anchors of contented involvement; 4) levels of thinking and performance; 5) strengthening the family as a resource for caregiving; and 6) review and integration of the previous sections.
  Interventions: Behavioral: PPA Tele-Savvy Pilot Intervention

INTERVENTIONS:
Behavioral: PPA Tele-Savvy Pilot Intervention — We will engage PPA caregivers in the process of adapting the existing Tele-Savvy program to fit their needs and then pilot test the adapted PPA Tele-Savvy program.

SUMMARY:
The primary goal of this pilot project is to adapt an evidence-informed on-line psychoeducation program (Tele-Savvy) to address the unique challenges facing informal caregivers of those living with PPA and geared toward achieving caregiver mastery in this population.

DETAILED DESCRIPTION:
The primary goal of this pilot project is to develop an evidence-informed on-line psychoeducation program (Tele-Savvy) based on the well-established Savvy Caregiver program to address the unique challenges facing informal caregivers of those living with Primary Progressive Aphasia (PPA) and to help these caregivers achieve mastery. Key elements of the adaptation process are to identify and adapt mechanistic elements of the Tele-Savvy intervention (increasing self-efficacy, mastery of new skills, increased knowledge of disease-specific symptoms and trajectories, problem-solving skills). We will engage PPA caregivers in the process of adapting the existing Tele-Savvy program to fit their needs and then pilot test the adapted PPA Tele-Savvy program.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

Informal (family or friends) caregivers of persons living with or deceased from PPA.

Age 18 or over Providing or have provided at least 2 hours per day of unpaid assistance, on average, for a person in the early-middle stage of PPA.

Must have access to a computer with adequate internet connection. Able to use a videoconferencing platform and receive email. Participants must be able to read, speak and understand English and have no uncorrectable vision or hearing deficits that might impede participation.

Aim 2:

Informal (family or friends) caregivers of persons living with PPA. Age 18 or over Providing at least 2 hours per day of unpaid assistance, on average, for a person in the early-middle stage of PPA.

Must have access to a computer with adequate internet connection. Able to use a videoconferencing platform and receive email. Must be able to read, speak and understand English and have no uncorrectable vision or hearing deficits that might impede participation.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Mastery Pearlin Caregiver Stress Scale Score | Baseline, 6-week follow-up
  Comprised of 6 domains from the full Pearlin Stress Scale. 1. Relational Deprivation: 6-24, higher scores indicate increased relational deprivation. 2. Role Captivity: 3 - 12, higher scores indicate an increased feeling of being trapped in the caregiver role. 3. Loss of Self: 2 - 8, higher scores indicate a greater loss of self. 4. Caregiving competence: 4 - 16, higher scores indicate greater caregiving competence. 5. Management of Situation: 4 - 16, higher scores indicate better management of the caregiving situation. 6. Management of Meaning: 9 - 36, higher scores indicate a better management of the meaning of the caregiving role.

SECONDARY OUTCOMES:
Change in Caregiver Depression Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, 6-week follow-up
  A 20-item scale that represents a symptom cluster consisting of negative affect, positive affect, interpersonal problems, and somatic activity based on feelings over the past week.Scores range 0 - 60. A score of 0-16 indicates little to no symptomatology, a score of 16 or more indicates depression with higher scores indicating increased severity.
Change in Caregiver Burden The Zarit Burden Interview score | Baseline, 6-week follow-up
  The interview was developed to measure subjective burden among caregivers of adults with dementia. The 22-item self-report inventory examines burden associated with functional/behavioral impairments and the home care situation. The items are worded subjectively, focusing on the affective response of the caregiver. Scores range 0 - 88. Lower scores indicate little to no burden. Higher scores indicate greater burden. A score of 17 or more is considered high burden.
Change in Caregiver Stress Perceived Stress Survey score | Baseline, 6-week follow-up
  This questionnaire is comprised of 10 items from the Perceived Stress Scale. Scores range 0 - 40. Higher scores indicating higher perceived stress. A score of 0-13 would be considered low stress. Scores from 14-26 would be considered moderate stress. Scores from 27-40 indicate high perceived stress.
Change in Positive Aspects of Caregiving (PCOS) Scale score | Baseline, 6-week follow-up
  Caregivers will be instructed that "In spite of all the difficulties involved in giving care to a family member with memory or health problems, good things can come out of caregiving experiences." The scale has 11 items, and overall scores range 0 - 44. Higher scores indicate a more positive view of the caregiving role while lower scores indicate less positive views of the caregiver role.
Change in Care recipient quality of life DEMQOL: Dementia Quality of Life Measure (Carer v4) score | Baseline, 6-week follow-up
  This 32 item questionnaire will be used to assess mood, cognitive status, and overall quality of life of the care recipient. Scores range 31 - 124. Lower scores indicate no subjective concerns about cognition or general health, while higher scores indicate a greater subjective concern about cognition and general health.
Change in Behavioral and Psychological Symptoms of Dementia Revised Memory and Behavior Problem Checklist (RMBPC) score | Baseline, 6-week follow-up
  This 24 item instrument measures the frequency of the care recipient's problem behaviors in the following domains: disruptive behavior (wandering, aggression), memory-related behavior (repeating questions and stories), and depression. Scores range 0 - 96 for frequency. Lower scores indicate little to no behavioral problems while higher scores indicate greater behavioral issues. Scores range 0 - 96 for reaction. Lower scores indicate little concern regarding the behavior on the part of the caregiver while higher scores indicate greater concern.

CONTACTS AND LOCATIONS:
Overall Officials: Darby Morhardt, PhD, Principal Investigator — Northwestern University; Darby Morhardt, PhD, Study Chair — Northwestern University; Darby Morhardt, PhD, Study Director — Northwestern University
Locations (1):
- Mesulam Center for Cognitive Neurology and Alzheimer's Disease, Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No